CLINICAL TRIAL: NCT06004427
Title: Investigation of the Effectiveness of Resistance Exercise Program Given With Diet in Obese Individuals.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, assistant professor, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar74
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Obesity
Keywords: resistant exercise; diet
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: resistance training (RT), (3 days/wk, 3 sets/day, 8-12 repetitions/set)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): regular diet program
  Interventions: Other: Diet program
- exercise group (Experimental): resistance exercise program
  Interventions: Other: Diet program; Other: Exercise training protocols

INTERVENTIONS:
Other: Diet program — A diet program will be prepared with the help of a dietitian at the beginning of 12 weeks for all participants who agree to participate in the study, and this program will be controlled by a dietitian once a month and completed at the end of 12 weeks.
Other: Exercise training protocols — calisthenic exercises exercises with lower and upper extremity theraband exercises with light dumbbells
  Arms: exercise group

SUMMARY:
The aim of this study is to examine the effects of diet and combined resistance exercise training on physical activity and sleep patterns compared to diet program alone.

DETAILED DESCRIPTION:
The study was planned as a randomized controlled trial. The groups will be divided into two as control group and exercise group by simple randomization method.While the normal diet program will be applied to the obese individuals in the control group, the individuals in the exercise group will be given resistance exercise training together with the diet program.Before and after the treatment, fatigue severity scale pittsburgh sleep quality scale international physical activity index questionnaires will be applied to the participants.In addition, sociodemographic characteristics and waist circumference measurement will be recorded. After the 12-week diet program, the data of the participants will be compared by making statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years or older.
* Having a Body Mass Index of 30 or higher.
* To have accepted the voluntary consent form that requires participation in the study.

Exclusion Criteria:

* Any neurological or psychological problems.
* Do not accept the voluntary consent form.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI) | 13 weeks
  The scale is a 19-item self-report scale that assesses sleep quality and impairment over the past month. It consists of 24 questions, 19 questions are self-report questions, 5 questions are questions to be answered by the spouse or roommate. The 18 scored questions of the scale consist of 7 components. Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficiency, Sleep Disorder, Sleeping Drug Use, and Daytime Dysfunction. Each component is evaluated over 0-3 points. The total score of the 7 components gives the scale total score. The total score ranges from 0 to 21. A total score greater than 5 indicates "poor sleep quality"
Fatigue Severity Scale (FSS) | 13 weeks
  There are 9 questions in the scale and each question consists of 7 points. The scale determines the fatigue status of individuals in the last 1 month. Questions are scored as Strongly disagree - Totally agree. The scale score is the average value of the questions. If the average score is 5 and above, it is considered as "fatigue".
International Physical Activity Questionnaire - Short Form | 13 weeks
  This questionnaire is a standardized tool for measuring physical activity, developed by researchers from various countries with the support of the World Health Organization (WHO) and Centers for Disease Control (CDC). Questionnaire, four areas of physical activity; It covers work, transportation, housework/gardening, and leisure activities, but also includes questions about time spent sitting as an indicator of inactivity. In each of the four areas, the energy expended in moderate and vigorous activities in the last 7 days, the number of days the activities were performed, and the number of activities performed during the day are recorded. The times are multiplied by the Metabolic Equivalent (MET) values per activity, and the results for all items are added to form the overall physical activity score. The question about sitting is not included in the physical activity score. Classification is made in three categories as physically inactive (3000 MET min/week).

CONTACTS AND LOCATIONS:
Overall Officials: Alara Livanur ÇELİK, Study Chair — Uskudar University
Locations (1):
- Üsküdar Unıversıty, Üsküdar, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Waters DL, Aguirre L, Gurney B, Sinacore DR, Fowler K, Gregori G, Armamento-Villareal R, Qualls C, Villareal DT. Effect of Aerobic or Resistance Exercise, or Both, on Intermuscular and Visceral Fat and Physical and Metabolic Function in Older Adults With Obesity While Dieting. J Gerontol A Biol Sci Med Sci. 2022 Jan 7;77(1):131-139. doi: 10.1093/gerona/glab111. PMID 33839788
- [Background] Dieli-Conwright CM, Courneya KS, Demark-Wahnefried W, Sami N, Lee K, Sweeney FC, Stewart C, Buchanan TA, Spicer D, Tripathy D, Bernstein L, Mortimer JE. Aerobic and resistance exercise improves physical fitness, bone health, and quality of life in overweight and obese breast cancer survivors: a randomized controlled trial. Breast Cancer Res. 2018 Oct 19;20(1):124. doi: 10.1186/s13058-018-1051-6. PMID 30340503
- [Background] Soriano-Maldonado A, Martinez-Forte S, Ferrer-Marquez M, Martinez-Rosales E, Hernandez-Martinez A, Carretero-Ruiz A, Villa-Gonzalez E, Barranco-Ruiz Y, Rodriguez-Perez MA, Torrente-Sanchez MJ, Carmona-Rodriguez L, Soriano-Maldonado P, Vargas-Hitos JA, Casimiro-Andujar AJ, Artero EG, Fernandez-Alonso AM. Physical Exercise following bariatric surgery in women with Morbid obesity: Study protocol clinical trial (SPIRIT compliant). Medicine (Baltimore). 2020 Mar;99(12):e19427. doi: 10.1097/MD.0000000000019427. PMID 32195937
- [Background] Villareal DT, Aguirre L, Gurney AB, Waters DL, Sinacore DR, Colombo E, Armamento-Villareal R, Qualls C. Aerobic or Resistance Exercise, or Both, in Dieting Obese Older Adults. N Engl J Med. 2017 May 18;376(20):1943-1955. doi: 10.1056/NEJMoa1616338. PMID 28514618
- [Background] Willis LH, Slentz CA, Bateman LA, Shields AT, Piner LW, Bales CW, Houmard JA, Kraus WE. Effects of aerobic and/or resistance training on body mass and fat mass in overweight or obese adults. J Appl Physiol (1985). 2012 Dec 15;113(12):1831-7. doi: 10.1152/japplphysiol.01370.2011. Epub 2012 Sep 27. PMID 23019316